CLINICAL TRIAL: NCT03856853
Title: A Phase III, Randomized, Double-blind, Placebo Controlled, Multicenter Clinical Trial to Evaluate the Efficacy and Safety of Pirfenidone in Subjects With Systemic Sclerosis-associated Interstitial Lung Disease (SSc-ILD)
Brief Title: Efficacy and Safety of Pirfenidone in Patient With Systemic Sclerosis-associated Interstitial Lung Disease
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Continent Pharmaceutical Co, Ltd. (Industry)
Collaborators: Shanghai Genomics, Inc. (Industry); GNI-EPS Pharmaceuticals, Inc. (GNI Group) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GNI-F647-1701
Record Dates: First submitted 2019-02-26; First posted 2019-02-27 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Systemic Sclerosis-associated Interstitial Lung Disease (Ssc-ild)
MeSH Terms: interventions — pirfenidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Experimental): pirfenidone group
  Interventions: Drug: Pirfenidone
- placebo group (Placebo Comparator): placebo group
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Pirfenidone — pirfenidone for SSc-ILD treatment
  Arms: treatment group
Other: placebo — as control
  Arms: placebo group

SUMMARY:
The purpose of this study is to evaluate the eEfficacy and safety of pirfenidone in subjects with systemic sclerosis-associated interstitial lung disease (SSc-ILD)

ELIGIBILITY:
Inclusion Criteria:

1.Female or male subjects aged between 18 and 75 years of age. 2.2013 ACR / EULAR classification criteria for SSc fulfilled. 3.SSc disease onset (defined by first non-Raynaud symptom) within 5 years. 4.SSc related Interstitial Lung Disease confirmed by HRCT. 5.Forced vital capacity (FVC) 40% to 70% predicted(include 40% and70% ). 6.Subject have the ability to understand and sign the informed consent before the trials.

Exclusion Criteria:

1. Subjects not fulfill all of the above inclusion criteria.
2. AST, ALT >1.5 x ULN.
3. Bilirubin >1.5 x ULN.
4. Creatinine clearance <30 mL/min.
5. Airway obstruction (pre-bronchodilator FEV1/FVC <0.7).
6. Other clinically significant pulmonary abnormalities.
7. Allergic to test drugs or components (e.g. lactose).
8. Clinical Significant Pulmonary hypertension:.

   1. Significant past clinical evidence or echocardiography of right heart failure.
   2. History of right heart catheterization showed that cardiac index ≤ 2 l/min/m2.
   3. Pulmonary hypertension, which needs to use EPoprostenol/ Treprostinil for parenteral treatment .
9. Cardiovascular diseases:

   1. Six weeks in severe hypertension, and out of control after treatment(≥160/100mmHg).
   2. Myocardial infarction within six months.
   3. A period of 6 months in unstable angina.
10. More than 3 digital fingertip ulcers or a history of severe digital necrosis requiring hospitalization or severe other ulcers.
11. Bleeding risk, including the following criterias:

    a. Predisposition to bleeding. b.Subjects need to the following treatments: i.Fibrinolysis, full-dose anticoagulation therapy(such as vitamin K antagonists, direct thrombin inhibitor, heparin, Hirudin ).

    ii. High dose antiplatelet therapy[Note: not prohibited to maintain equipment needed indwelling venous pathway prophylactic low dose of heparin or heparin fluid (e.g. enoxaparin, daily 4000 I.U. s.c.) and the prevention of the use of antiplatelet therapy (e.g. acetylsalicylic acid, until 325 mg/d, or other antiplatelet dose of 75 mg/d the same dose of clopidogrel, or treatment)].

    c.history of hemorrhagic central nervous system (CNS) event within last year. d. Any of the following conditions within 3 months: i.Hemoptysis or hematuria ii. Active gastrointestinal bleeding or gastrointestinal ulcer. iii. major trauma or major surgery (researchers determined). e.coagulation parameters:international normalised ratio (INR) >2, prolongation of prothrombin time (PT) and partial thromboplastin time (PTT) by >1.5 x ULN)
12. May interfere with detection procedures (such as interrupt oxygen intolerance in pulmonary function tests) or based on the researchers estimate, may affect the test to participate in or participate in the test may put patients at risk of disease or other complications (such as caused by SSc severe gastrointestinal symptoms).
13. Researchers determined that life expectancy was due to other diseases (non SSc) for a period of up to 2.5 years.
14. Clinical signs of malabsorption or needing parenteral nutrition.
15. History of thrombotic event within last year(Including stroke and transient ischemic attack).
16. Previous treatment with nintedanib or pirfenidone.
17. Use the following medicine:

    1. Treatment with prednisone >10 mg/day within 2 weeks.
    2. Treatment with azathioprine, hydroxychloroquine, colchizine, D-penicillamine, sulfasalazine within 8 weeks .
    3. Treatment with cyclophosphamide, rituximab, tocilizumab, abatacept, leflunomide, tacrolimus, newer anti-arthritic treatments like tofacitinib and ciclosporine A, potassium para-aminobenzoate within 6 months.
18. Unstable background therapy with cyclophosphamide or mycophenolate mofetil / sodium or methotrexate (not allow treatment). Patients must or A. patients cannot receive immunosuppressive therapy, sodium cyclophosphamide or mycophenolate mofetil / or MTX stable or B. within 6 months of acceptance, and in at least 6 months after randomization, the treatment to keep the background stable (exclusion criteria 16 and 17 and the combined use of early precautions).
19. Previous or planned hematopoietic stem cell transplantation next year.
20. Major surgery is planned during the treatment period.
21. Pregnancy or lactation or make a schedule during the trials.
22. Give the drug 28 days before or after administration of the 3 month period, women of childbearing age * are unwilling or unable to use contraceptive methods highly effective (according to ICH M3 (R2)), a highly effective means in the correct and consistent application of a barrier method when the failure rate of less than 1% per year. * women of childbearing age is defined has undergone menarche and in line with "infertile women" standard "[female infertile women" is defined as: postmenopausal period (12 months without menstruation, no other medical reasons) or permanent sterilization (e.g., tubal occlusion, hysterectomy, bilateral ovarian resection or bilateral tubal resection women)].

(23)According to the researchers,exhibited evidence of alcohol or drug abuse. (24)Patients who were unable to understand or comply with the procedure were included in the self-administered questionnaire, which was completed without help.

25.Patients with underlying chronic liver disease (Child Pugh A, B, C hepatic impairment).

26.Clinical signs of malabsorption or needing parenteral nutrition. 27.With active peptic ulcer. 28.With mental illness . 29.Within 3 months to participate in other clinical trials. 30.Researchers determined that they did not participate in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2018-06-15 (Actual); Primary Completion 2021-02-10 (Estimated); Study Completion 2021-05-10 (Estimated)

PRIMARY OUTCOMES:
Relative change from baseline (%) of FVC% | 52 Weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Zhang, Ling, Beijing, Beijing Municipality, China